CLINICAL TRIAL: NCT00818155
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Desvenlafaxine Succinate Sustained Release Administered Orally to Healthy Chinese Subjects.
Brief Title: Study Evaluating the Safety, Tolerability and Pharmacokinetics of Desvenlafaxine Succinate SR in Healthy Chinese Male and Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A1-197; B2061064 (Other: Pfizer)
Record Dates: First submitted 2008-12-23; First posted 2009-01-07 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- desvenlafaxine succinate SR (Experimental): desvenlafaxine succinate SR
  Interventions: Drug: desvenlafaxine succinate SR
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: desvenlafaxine succinate SR — desvenlafaxine succinate SR
  Arms: desvenlafaxine succinate SR
Other: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of desvenlafaxine succinate SR in healthy male and female Chinese subjects. The amount of drug in the body and the effects of the drug will also be evaluated.

ELIGIBILITY:
Inclusion:

1. Men or non-pregnant, non-lactating women, 18 to 45 years of age inclusive on study day 1.
2. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG)
3. Nonsmoker or smoker of fewer than 10 cigarettes (half a pack) a day.

Exclusion:

1. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.
2. History of epilepsy or seizure disorder (except history of a single childhood febrile seizure).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as evaluated from reported adverse events, scheduled physical examinations, vital sign measurements, cardiac rhythm monitoring, 12 lead ECG and clinical laboratory results. | 2 months

SECONDARY OUTCOMES:
Pharmacokinetics as evaluated from blood and urine concentrations of desvenlafaxine | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer